CLINICAL TRIAL: NCT00758199
Title: Determination of Optimum Duration of Treatment With Bromfenac (Xibrom) Eyedrops Following Cataract Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bp Consulting, Inc (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008-0036
Record Dates: First submitted 2008-09-22; First posted 2008-09-25 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Cataracts
MeSH Terms: conditions — Cataract | interventions — bromfenac; Moxifloxacin; prednisolone acetate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 2 (Active Comparator): Moxifloxacin
  Interventions: Drug: Moxifloxacin hydrochloride
- 3 (Placebo Comparator): Prednisolone Acetate
  Interventions: Drug: Prednisolone Acetate
- 1 (Active Comparator): Bromfenac
  Interventions: Drug: Bromfenac

INTERVENTIONS:
Drug: Bromfenac — Group 1: Bromfenac BID for 3 weeks Group 2: Bromfenac BID for 6 weeks
  Other Names: Bromfenac (Xibrom)
  Arms: 1
Drug: Moxifloxacin hydrochloride — Group 1 and Group 2:Moxifloxacin hydrochloride 1 day prior to surgery-continue for six days after surgery.
  Other Names: Moxifloxacin hydrochloride (Vigamox)
  Arms: 2
Drug: Prednisolone Acetate — Group 1 and Group 2:Prednisolone Acetate for 3 weeks in a tapering schedule (week 1: TID; week 2: BID, week 3:QD).
  Other Names: Omni-Pred
  Arms: 3

SUMMARY:
The objective of this study is to determine if an extension of bromfenac BID monotherapy is effective in the decreasing retinal thickening post cataract IOL placement surgery. No studies exist on how long to treat with an NSAID post cataract IOL placement surgery. Currently, NSAID therapy post IOL placement surgery is in conjunction with steroid treatment, lasting approximately 3 weeks. This study is designed to examine if there is benefit to extending NSAID monotherapy in regards to macular thickening and the incidence of CME.

ELIGIBILITY:
Inclusion Criteria:

* Male or female >18 years of age scheduled to undergo bilateral cataract surgery
* Patients with systemic diseases will be enrolled only if there are no ocular manifestations of their disease (e.g. diabetics with normal retinal exams)
* Expected visual outcome of BCVA > [greater than or equal to] 20/30 postoperatively
* Ability to provide informed consent, take study medications as directed, and likely to complete all study visits

Exclusion Criteria:

* Known contraindication to any study medication or any of their components
* Required use of ocular medications other than the study medications during the study
* Significant AMD, epi-retinal membrane, retinal vein occlusion, diabetic macular edema, or any macular disease predisposing them to cystoid macular edema.
* Posterior capsule rupture, Vitreous loss during surgery or any other complication that in the surgeon's opinion, could reduce potential for targeted visual outcome
* Anticipated need for mechanical iris dilating devices

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2008-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
OCT with macular thickening | 3-6 weeks

SECONDARY OUTCOMES:
Incidence of CME | 3-6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Altos Eye Physicians, Los Altos, California, United States